CLINICAL TRIAL: NCT04855396
Title: The Biomarkers in the Hyperbaric Oxygen Brain Injury Treatment Trial (BioHOBIT)
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Frederick Korley, MD, PhD, Associate Professor of Emergency Medicine, University of Michigan
Other Study IDs: Pro00024234
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury
Keywords: Monitoring Biomarkers; Predictive Biomarkers; Glial Fibrillary Acidic Protein; Neurofilament Light Chain; High Sensitivity C-Reactive Protein
MeSH Terms: conditions — Brain Injuries, Traumatic; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum/plasma and CSF samples will be analysed for measurments of: Glial fibrillary acidic protein (GFAP), neurofilament light chain (NfL) and high sensitivity c-reactive protein (hsCRP)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Severe Traumatic Brain Injury: Participants will be enrolled in the HOBIT trial

SUMMARY:
There are no therapeutic agents that have been shown to improve outcomes from severe traumatic brain injury (TBI). Critical barriers to progress in developing treatments for severe TBI are the lack of: 1) monitoring biomarkers for assessing individual patient response to treatment; 2) predictive biomarkers for identifying patients likely to benefit from a promising intervention. Currently, clinical examination remains the fundamental tool for monitoring severe TBI patients and for subject selection in clinical trials. However, these patients are typically intubated and sedated, limiting the utility of clinical examinations. Validated monitoring and predictive biomarkers will allow titration of the dose of promising therapeutics to individual subject response, as well as make clinical trials more efficient by enabling the enrollment of subjects likely to benefit. Glial fibrillary acidic protein (GFAP), neurofilament light chain (NfL) and high sensitivity c-reactive protein (hsCRP) are promising biomarkers that may be useful as 1) monitoring biomarkers; 2) predictive biomarkers in severe TBI trials. Although the biological rationale supporting their use is strong, significant knowledge gaps remain. To address these gaps in knowledge, we propose an ancillary observational study leveraging an ongoing severe TBI clinical trial that is not funded to collect biospecimen. The Hyperbaric Oxygen in Brain Injury Treatment (HOBIT) trial, a phase II randomized control clinical trial that seeks to determine the dose of hyperbaric oxygen therapy (HBOT) that that has the highest likelihood of demonstrating efficacy in a phase III trial. The proposed study will: 1) validate the accuracy of candidate monitoring biomarkers for predicting clinical outcome; 2) determine the treatment effect of different doses of HBOT on candidate monitoring biomarkers; and 3) determine whether there is a biomarker defined subset of severe TBI that responds favorably to HBOT. This proposal will: 1) inform a go/no-go decision for a phase III trial of HBOT by providing adjunctive evidence of the effect of HBOT on key biological pathways through which HBOT is hypothesized to affect outcome; 2) provide evidence to support further study of the first monitoring biomarkers of severe TBI; 3) increase the likelihood of success of a phase III trial by identifying the sub-population of severe TBI likely to benefit from HBOT; 4) create a repository of TBI biospecimen which may be accessed by other investigators.

This study is related to NCT04565119

DETAILED DESCRIPTION:
The Investigators will obtain an initial set of biospecimens (serum, plasma, CSF, DNA) as soon as feasible after randomization to a HOBIT study arm, but no later than 24 hours from injury. Subsequent biospecimens will be obtained every 8 hours (+/- 1 hour) for the first 24 hours post-enrollment. This will allow the characterization of acute changes in biomarker levels. On study days 2, 3, 5, 7 and 14 biospecimens will be obtained once a day to allow characterization of sub-acute changes in biomarker levels. If feasible, samples should be collected at 8am (+/- 2 hours) to minimize the effects of circadian rhythm on biomarker levels. In addition, during the first 5 days of the study, one set of biospecimen will be collected 4 hours after HBO treatment to examine the acute effects of HBO treatment on biomarkers. This will not apply to those randomized to non-HBOT groups. During the 6-month visit, 1 tablespoon (15 ml) of blood will be collected. In addition, for subjects who have an external ventricular drain in place, 5 cc of CSF will be collected at each time point if feasible. Since subjects are unlikely to have an EVD after the first week post-injury, CSF samples will be collected only for as long as the EVD is in place.

BioHOBIT will utilize data collected in the HOBIT trial. This data includes: demographic data and clinical data such as injury characteristics, vital signs, head CT findings, laboratory data and data on physiologic parameters such as intracranial pressure (ICP), partial pressure of brain tissue oxygen (PbtO2), mean arterial pressure (MAP), and cerebral perfusion pressure (CPP), among others.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in HOBIT (this is an ancillary study to the HOBIT Trial)

Exclusion Criteria:

* Profoundly anemic (subjects who are profoundly anemic require blood transfusion)
* Blood samples cannot be obtained

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators plan to enroll a maximum of 150 male and female subjects among multiple clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Unfavorable Neurologic Outcome | 6-months post injury
  Glasgow Outcome Scale Extended with a score of <5. Score ranges from 1 to 8, with 1 = death, 8 = Complete Recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Korley, MD, PhD, Principal Investigator — University of Michigan; William Barsan, MD, Principal Investigator — University of Michigan; Gaylan Rockswold, MD, PhD, Principal Investigator — Hennepin Healthcare; Byron Gajewski, PhD, Principal Investigator — University of Kansas
Locations (11):
- United States (10):
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - St. Mary's Medical Center, West Palm Beach, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Detroit Receiving Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Hospital, Durham, North Carolina
  - OSU Wexner Medical Center, Columbus, Ohio
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No